CLINICAL TRIAL: NCT04457154
Title: Inspire Pediatric Post-Approval Registry
Brief Title: Pediatric Post-Approval Registry
Status: Recruiting | Type: Observational
Sponsor: Inspire Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-002
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-08

CONDITIONS: Obstructive Sleep Apnea
Keywords: Pediatric; Apnea-hypopnea Index; Sleep Breathing Disorders
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Pediatric Postmarket Surveillance: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Registry Population: Pediatric subjects (age 18-21 years) who are undergoing implant of the Inspire Upper Airway Stimulation System for the treatment of moderate to severe obstructive sleep apnea (OSA)
  Interventions: Device: Inspire Upper Airway Stimulation System

INTERVENTIONS:
Device: Inspire Upper Airway Stimulation System — Implant of the Inspire Upper Airway Stimulation System

SUMMARY:
This registry is a prospective, multi-center, single-arm study of pediatric subjects (ages 18-21 years) who are undergoing implant of the Inspire Upper Airway Stimulation (UAS) System for the treatment of moderate or severe obstructive sleep apnea (OSA). Implanted subjects will be followed for 5 years post-implant.

DETAILED DESCRIPTION:
This registry is a prospective, multi-center, single-arm study of pediatric subjects (ages 18-21 years) who are undergoing implant of the Inspire Upper Airway Stimulation (UAS) System for the treatment of moderate or severe obstructive sleep apnea (OSA). Implanted subjects will be followed for 5 years post-implant.

Subjects will be recruited in accordance with the approved Inspire UAS indication for use and will only include those subjects who are within the new age indication (18-21 years of age). Implanted subjects must meet the registry eligibility criteria. Those subjects that are enrolled but fail to meet the eligibility criteria will be considered screen failures.

This registry will collect safety and effectiveness data on 60 implanted subjects at a minimum of 5 qualified clinical centers in the United States.

Study data will be collected at the following timepoints:

Baseline (pre-implant) Implant Activation (1 month post-implant) 6 Months post-implant

1, 2, 3, 4, 5 years post-implant

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 18 and 21 years of age;
2. Subject has a diagnosis of moderate to severe OSA (15 ≤ AHI ≤ 65) based on a recent sleep study;
3. Subject has documented failure of, or intolerance to, positive airway pressure treatments, despite attempts to improve compliance;
4. Subject is contraindicated for, or not effectively treated by, adenotonsillectomy;
5. Subject has followed standard of care in considering all other alternative/adjunct therapies;
6. Subject is willing and able to have stimulation hardware permanently implanted and to use the patient remote to activate the stimulation;
7. Subject is willing and able to return for follow-up visits, undergo sleep studies (including in-lab and at-home), and complete questionnaires related to the registry;
8. Subject is willing and able to provide informed consent.

Exclusion Criteria:

1. Subject has a combination of central + mixed apneas > 25% of the total apnea-hypopnea index (AHI);
2. Subject has any anatomical finding that would compromise the performance of upper airway stimulation, such as the presence of complete concentric collapse of the soft palate;
3. Subject has any condition or procedure that has compromised neurological control of the upper airway;
4. Subject is unable, or does not have the necessary assistance, to operate the patient remote;
5. Subject is pregnant or plans to become pregnant;
6. Subject has an implantable device that may be susceptible to unintended interaction with the Inspire System;
7. Subject has a terminal illness with life expectancy < 12 months;
8. Any other reason the investigator deems the subject is unfit for participation in the registry.

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pediatric subjects (ages 18-21 years) who are undergoing implant of the Inspire Upper Airway Stimulation (UAS) System for the treatment of moderate or severe obstructive sleep apnea (OSA).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of device and/or procedure related adverse events over time | Implant through 5 years post-implant
  relevant adverse events will be collected and reported
Evaluation of the improvement of Apnea Hypopnea Index (AHI) over time | through 5 years post-implant
  Baseline (pre-implant) AHI compared to AHI after implant (collected and reported at annual study visits). The Apnea Hypopnea Index (AHI) is the number of apnea and hypopnea events per hour of sleep. A lower AHI indicates less severe sleep apnea.

SECONDARY OUTCOMES:
Evaluation of improvement in Oxygen Desaturation Index (ODI) over time | through 5 years post-implant
  Baseline (pre-implant) Oxygen Desaturation Index (ODI) compared to ODI after implant (collected and reported at annual study visits). The Oxygen Desaturation Index (ODI) is the number of oxygen desaturations, with at least a 4% drop from baseline, per hour. A lower ODI indicates less severe sleep apnea.
Evaluation of improvement in T90 (defined as total sleep time spent with arterial oxygen saturation (SaO2) < 90%) over time | through 5 years post-implant
  Baseline (pre-implant) T90 compared to T90 after implant (collected and reported at annual study visits). T90 is defined as the total sleep time spent with arterial oxygen saturation (SaO2) < 90%. A lower T90 indicates less severe sleep apnea.
Evaluation of improvement of Epworth Sleepiness Scale (ESS) over time | through 5 years post-implant
  Baseline (pre-implant) Epworth Sleepiness Scale (ESS) compared to ESS after implant (collected and reported at annual study visits). The Epworth Sleepiness Scale is a validated, self-report instrument that rates a subject's tendency to fall asleep in eight common daily situations. Scores range from 0 to 24, with a lower score indicating less daytime sleepiness. An ESS score of 10 or less is equivalent to the normalized population.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Childrens Hospital of Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Duke University, Durham, North Carolina
  - Cincinnati Childrens Hospital, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Sewickley, Pennsylvania
  - University of Texas Southwestern/Children's Hospital of Dallas, Dallas, Texas
  - Children's Hospital of the King's Daughters/East Virginia Medical School, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Undecided